CLINICAL TRIAL: NCT05986786
Title: Single-arm, Open Label, Multicenter Clinical Study to Evaluate the Handling and Safety of AVT06 Pre-filled Syringe (PFS) in Subjects With Chorioretinal Vascular Disease Followed by an Optional Extension Phase of AVT06 Pre-filled Syringe (PFS)
Brief Title: Clinical Study to Evaluate the Handling and Safety of AVT06 PFS in Subjects With Chorioretinal Vascular Disease
Acronym: ALVOEYE-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVT06-GL-D01
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Chorioretinal Vascular Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVT06 (proposed aflibercept biosimilar) PFS (Experimental): IVT injection with a PFS containing the proposed aflibercept biosimilar AVT06
  Interventions: Device: Patients will receive 1 IVT injection of AVT06 PFS depending on their chorioretinal vascular disease schedule

INTERVENTIONS:
Device: Patients will receive 1 IVT injection of AVT06 PFS depending on their chorioretinal vascular disease schedule — Patient will receive AVT06 (proposed aflibercept biosimilar) PFS injection

SUMMARY:
This is a single-arm, open label, multicenter clinical study to evaluate the handling and safety of AVT06 pre-filled syringe (PFS) in subjects with chorioretinal vascular disease followed by an optional extension phase of AVT06 pre-filled syringe (PFS)

ELIGIBILITY:
Inclusion Criteria :

* Male or female ≥18 years old
* Subjects with diagnosis of nAMD (wet), DME, RVO, DR, or myopic CNV in the study eye
* Study eye considered by the Principal Investigator to be indicated for treatment with aflibercept
* Subjects must sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form (ICF) before any study-specific procedures
* Willing and able to comply with all study procedures and be likely to complete the study
* Subjects must be able to follow the contraception requirements

Exclusion Criteria (selected):

* Any concurrent ocular condition in the study eye which, in the opinion of the Principal Investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of IVT injections, or which otherwise may interfere with the injection procedure or with evaluation of safety
* Current systemic infectious disease or a therapy for active infectious disease Any condition that, in the Principal Investigator's opinion, can interfere with full participation in the study, including administration of the study treatment and attending required visits; can pose a significant risk to the subject, or interfere with interpretation of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Proportion of AVT06 injections successfully administered with PFS at Day 1 to demonstrate effective and safe handling of AVT06 PFS. | Day 1
  Proportion of AVT06 injections successfully administered with PFS at Day 1
Incidence of ocular TEAEs, AESIs, and SAEs on the study eye from Baseline to Week 4 to evaluate ocular safety of AVT06 delivered from the PFS | Week 4
  Incidence of ocular TEAEs, AESIs, and SAEs on the study eye from Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Juergen Agostini, Principal Investigator — University Clinic Freiburg
Locations (1):
- 4001, Tbilisi, Georgia